CLINICAL TRIAL: NCT06850454
Title: A Prospective Randomized, Double-blind Controlled Trial of Olanzapine Versus Placebo in Addition to Ondansetron Plus Dexamethasone As Antiemetic Prophylaxis in Patients Receiving Moderately Emetogenic Chemotherapy
Brief Title: Olanzapine Versus Placebo for Moderately Emetogenic Chemotherapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, suthinee ithimakin, Associate professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 811/2567(IRB3)
Record Dates: First submitted 2024-11-07; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-11

CONDITIONS: Chemotherapy Induced Nausea and Vomiting
Keywords: olanzapine; moderately emetogenic chemotherapy; carboplatin; irinotecan; oxaliplatin
MeSH Terms: conditions — Vomiting | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- olanzapine (Experimental): olanzapine 5 mg on day 1-4
  Interventions: Drug: olanzapine
- placebo (Placebo Comparator): placebo 5 mg day 1-4
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: olanzapine — olanzapine 5 mg oral prior to chemotherapy on day 1 and daily on day 2-4
  Arms: olanzapine
Drug: Placebo — placebo 5 mg oral prior to chemotherapy on day 1 and daily on day 2-4
  Arms: placebo

SUMMARY:
A study comparing efficacy of olanzapine versus placebo to prevent nausea and vomiting from moderate emetic risk chemotherapy

DETAILED DESCRIPTION:
A randomized study comparing olanzapine versus placebo in addition to standard antiemetic regimen for preventing nausea and vomiting from moderately emetogenic chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed cancer patients who will be started on first dose of oxaliplatin, irinotecan or carboplatin
* age of >18 years old

Exclusion Criteria:

* pregnancy or breast feeding
* has emetic episode within 24 hours
* gut obstruction
* uncontrolled brain metastasis
* allergy to or current use of olanzapine
* concomittant moderate or high emetogenic chemotherapy on day 2-5
* Total bilirubin > 2 mg/dl or creatinine clearance < 30 ml/min
* unable to swallow drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
total protection rate of nausea and vomiting | 5 days
  Proportion of patients without vomiting or requiring rescue therapy and VAS nausea score of less than 25 mm

SECONDARY OUTCOMES:
no nausea rate | 5 days
severity of nausea and vomiting | 5 days
  Number of patients with grade of nausea or vomiting according to CT-CAE
adverse events | 5 days
  Number of patients with other adverse event(s)
rescue therapy | 5 days
  Number of patients requiring additional therapy
quality of life score | 5 days
  EQ-5D-5L score
Cost | 5 days
  medical cost excluding chemotherapy and prophylactic measures

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon request
Supporting Information: Study Protocol, CSR
Time Frame: After study completion and published, lasting for 5 years
Access Criteria: The IPD will be provided upon request by email.

REFERENCES:
- [Background] Shen J, Zhao J, Jin G, Li H, Jiang Y, Wu Y, Gao J, Chen F, Li J, Wang W, Li Q. A prospective randomized controlled clinical trial investigating the efficacy of low-dose olanzapine in preventing nausea and vomiting associated with oxaliplatin-based and irinotecan-based chemotherapy. J Cancer Res Clin Oncol. 2024 May 28;150(5):283. doi: 10.1007/s00432-024-05712-7. PMID 38806870
- [Background] Yamamoto S, Iihara H, Uozumi R, Kawazoe H, Tanaka K, Fujita Y, Abe M, Imai H, Karayama M, Hayasaki Y, Hirose C, Suda T, Nakamura K, Suzuki A, Ohno Y, Morishige KI, Inui N. Efficacy and safety of 5 mg olanzapine for nausea and vomiting management in cancer patients receiving carboplatin: integrated study of three prospective multicenter phase II trials. BMC Cancer. 2021 Jul 19;21(1):832. doi: 10.1186/s12885-021-08572-3. PMID 34281514